CLINICAL TRIAL: NCT01343355
Title: Open-Label, Exploratory Study of the Efficacy and Safety of Tamibarotene(AM80H) for HTLV-1 Associated Myelopathy/ Tropical Spastic Paraparesis (HAM/TSP)
Brief Title: Efficacy and Safety of Tamibarotene(AM80H) for HTLV-1 Associated Myelopathy/ Tropical Spastic Paraparesis (HAM/TSP)
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: St. Marianna University School of Medicine (Other)
Responsible Party: Yoshihisa Yamano, MD, associate professor, Department of Molecular Medical Science, Institute of Medical Science
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AM80H-01
Record Dates: First submitted 2011-04-25; First posted 2011-04-28 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-07

CONDITIONS: HTLV-I-Associated Myelopathy
Keywords: Tropical Spastic Paraparesis; HAM; TSP
MeSH Terms: conditions — Paraparesis, Tropical Spastic | interventions — tamibarotene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Tamibarotene — Oral administration of tamibarotene 2 mg daily over a period of 12 weeks, then 4mg daily for another 12 weeks.

SUMMARY:
An open-label, non-randomised, uncontrolled, proof-of-concept study of patients with HTLV-I-associated myelopathy/Tropical Spastic Paraparesis (HAM/TSP). Participants will receive oral administration of tamibarotene in the amount of 2 mg daily over a period of 12 weeks, then 4mg daily for another 12 weeks. The patients will be followed up for further 8 weeks. Efficacy will be monitored by measuring clinical scores including motor and urination function, HTLV-1 proviral load, immunological parameters, and markers in the spinal fluid. Safety will be evaluated at the same time.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been diagnosed as HAM according to the WHO criteria
* Patients who are positive for HTLV-I antibody in the spinal fluid
* Patients, if female, who are not pregnant or breastfeeding, either agreed to take contraceptive measures during and two years after the treatment, or sterile
* Patients, if male, who agreed to take contraceptive measures during and six months after the treatment
* Patients who have been informed and understood the contents of the study and consented to participate in the signed form.

Exclusion Criteria:

* Patients who has a rapid progress in the symptoms defined as an increase of two or more in Osame's Motor Disability Score for HAM patients in the past one year.
* Patients of hyperlipidemia (serum triglyceride higher than 400 mg/dL)
* Patients who were administered new or increased dose of corticosteroid in the past 8 weeks before the intervention
* Patients who received steroid pulse therapy in the past 8 weeks before the intervention
* Patients who were administered new or increased dose of immunosuppressant in the past 8 weeks before the intervention
* Patients with a history of serious drug allergy
* Patients with significant complication such as malignancy, severe heart failure, and other serious diseases.
* Patients who were in the past administered etretinate.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-03 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Change in Soluble IL-2 Receptor level in peripheral blood | 0, 4, 8, 12, 16, 20, 24, 28 and 32 weeks
Change in HTLV-I viral load in peripheral blood | 0, 4, 8, 12, 16, 20, 24, 28 and 32 weeks
Change in T cell population in peripheral blood | 0,12, 24, 28 and 32 weeks
Change in cerebrospinal fluid examination | baseline and after the treatment defined as from 24 to 32 weeks

SECONDARY OUTCOMES:
Change in Osame's Motor Disability Score for HAM patients | 0, 4, 8, 12, 16, 20, 24, 28 and 32 weeks
Change in The Expanded Disability Status Scale (EDSS) | 0, 4, 8, 12, 16, 20, 24, 28 and 32 weeks
Change in timed 10m walk | 0, 4, 8, 12, 16, 20, 24, 28 and 32 weeks
Change in Manual Muscle Testing and vibratory perception of the lower limbs | 0, 4, 8, 12, 16, 20, 24, 28 and 32 weeks
Change in Modified Ashworth Scale | 0, 4, 8, 12, 16, 20, 24, 28 and 32 weeks
Change in Urination function and defecation score | 0, 4, 8, 12, 16, 20, 24, 28 and 32 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yoshihisa Yamano, MD, Principal Investigator — St. Marianna University School of Medicine
Locations (1):
- Iseikai Medical Corporation, Shoyo Kashiwadai Hospital, Kanagawa, Japan